CLINICAL TRIAL: NCT06125951
Title: A Phase 2b/3, Double-Blind, Placebo-Controlled, Parallel-Group, 36-Week, 2-Arm Trial to Assess the Safety, Tolerability, and Efficacy of Xanamem® 10 mg Daily in Patients With Mild or Moderate Dementia Due to Alzheimer's Disease
Brief Title: Effect of 10 mg Xanamem on Dementia Due to Alzheimer's Disease
Acronym: XanaMIA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Actinogen Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACW0009
Record Dates: First submitted 2023-10-23; First posted 2023-11-09 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Dementia Moderate; Dementia, Mild; Alzheimer Disease
Keywords: Xanamem; Actinogen; Alzheimer's Disease; Cortisol; emestedastat
MeSH Terms: conditions — Dementia; Lymphoma, Follicular; Alzheimer Disease | interventions — UE2343

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 10 mg Xanamem (Experimental): 10 mg Xanamem tablet, to be administered orally once every morning with or without food
  Interventions: Drug: Xanamem
- Placebo (Placebo Comparator): Placebo tablet, to be administered orally once every morning with or without food
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xanamem — Xanamem drug product is formulated as an immediate-release film-coated tablet formulation for oral administration. Each Xanamem tablet contains 10 mg Xanamem (UE2343) drug substance and excipients.
  Other Names: UE2343
  Arms: 10 mg Xanamem
Drug: Placebo — Matching placebo which is identical in appearance to the test product (10 mg Xanamem once daily) except that it contains no active ingredient.
  Arms: Placebo

SUMMARY:
Xanamem® is being developed as a potential treatment for symptomatic, early stages of Alzheimer's Disease (AD) and Major Depressive Disorder (MDD).

This XanaMIA Phase 2b/3 study is to investigate the safety, tolerability, and efficacy of Xanamem in in mild or moderate dementia due to AD. Trial participants will be randomized to either receive 10mg of Xanamem once daily or a placebo for 36 weeks at a 1:1 ratio in a double-blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 50 years or older, inclusive at the time of Screening.
* Clinical syndrome of mild or moderate dementia, likely to be due to AD in the opinion of the Investigator, at Screening, including meeting the following criteria:

  1. Clinical Dementia Rating (CDR) global score of 0.5 to 1.0
  2. Mini-mental state examination (MMSE) score of 18 to 26
  3. Magnetic resonance imaging (MRI) or computerized tomography (CT) scan within 1 year prior to randomization that excludes alternative diagnoses for dementia such as large stroke, likely vascular dementia, brain tumor, subdural hematoma, or other non-AD dementia type findings
  4. Positive plasma AD biomarker signature at Pre-screening, comprising fasting levels of a tau species protein.
* If receiving symptomatic AD medications, the dosing regimen must have been stable for 3 months prior to Screening.
* Has a consenting trial partner who, in the Investigator's judgment, has frequent and sufficient contact with the participant to be able to provide accurate information as to the participant's cognitive and functional abilities. The trial partner must be available to provide information to the Investigator and trial site staff about the participant and agrees to attend all trial site visits in person for scale completion. A trial partner should be available for the duration of the trial. The measure of adequate availability will be at the Investigator's discretion.
* Participants must be able to comfortably abstain from caffeine intake for 4 hours prior to scheduled cognitive assessments.
* Smokers are eligible if they are able to comfortably abstain from nicotine / tobacco products for 2 hours prior to scheduled cognitive assessments.
* Must provide written informed consent to participate in the trial and be willing and able to participate for the maximum of 9 months of treatment and up to 11.5 months of site visits.

Exclusion Criteria:

* Use of anti-amyloid or anti-tau antibody within 6 months.
* Diagnosis of a non-AD dementia including traumatic brain injury.
* Diagnosis of an active major mental illness of concern in the opinion in the Investigator, including major depressive disorder, bipolar illness, or schizophrenia.
* Participation in another clinical trial of a drug or device
* Has a body mass index or body weight that will interfere with participation in the trial, including inadequate venous access to complete the trial assessments, to be determined at the discretion of the Investigator.
* Previous clinically significant systemic illness or infection, including test positive COVID-19, within the past 4 weeks prior to Screening.
* Clinical diagnosis of Type I or Type II diabetes requiring insulin.
* Exhibit physical, cognitive, or language impairments, in the opinion of the Investigator, of such severity as to adversely affect the validity of the data derived from the neuropsychological tests.
* Trial participants with evidence of current infection with HIV, hepatitis B, or hepatitis C.
* Participants with a history of clinically significant drug abuse or addiction in the past 2 years
* Evidence or history of alcohol abuse

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Effects of 10 mg Xanamem on integrated cognitive and functional abilities | 36 weeks
  Change from Baseline to end of treatment (EOT) in the Clinical Dementia Ratio - Sum of Boxes (CDR-SB). The CDR-SB is calculated as an average score, with lower scores indicating improvement.
Incidence and severity of treatment-emergent adverse events (TEAEs) [safety and tolerability of Xanamem] | 36 weeks
  Incidence and severity of TEAEs

CONTACTS AND LOCATIONS:
Overall Officials: Global Program Lead, Study Director — Actinogen Medical Ltd
Locations (35):
- United States (20):
  - ACW Investigative Site 218, Carlsbad, California
  - ACW Investigative Site 213, Orange, California
  - ACW Investigative Site 209, Sherman Oaks, California
  - ACW Investigative Site 211, Denver, Colorado
  - ACW Investigative Site 208, Englewood, Colorado
  - ACW Investigative Site 203, Delray Beach, Florida
  - ACW Investigative site 201, Miami, Florida
  - ACW Investigative site 202, New Port Richey, Florida
  - ACW Investigative site 204, Orlando, Florida
  - ACW Investigative site 205, The Villages, Florida
  - ACW Investigative Site 207, Decatur, Georgia
  - ACW Investigative Site 206, Toms River, New Jersey
  - ACW Investigative Site 214, Albany, New York
  - ACW Investigative Site 219, Staten Island, New York
  - ACW Investigative Site 210, Dayton, Ohio
  - ACW Investigative Site 217, Independence, Ohio
  - ACW Investigative Site 212, Portland, Oregon
  - ACW Investigative Site 216, East Providence, Rhode Island
  - ACW Investigative Site 220, Austin, Texas
  - ACW Investigative Site 215, Bellevue, Washington
- Australia (15):
  - ACW Investigative Site 106, Darlinghurst, New South Wales
  - ACW Investigative Site 103, Erina, New South Wales
  - ACW Investigative Site 102, Kogarah, New South Wales
  - ACW Investigative Site 107, Macquarie Park, New South Wales
  - ACW Investigative Site 111, Newcastle, New South Wales
  - ACW Investigative Site 113, Birtinya, Queensland
  - ACW Investigative Site 105, Chermside, Queensland
  - ACW Investigative Site 114, Bedford Park, South Australia
  - ACW Investigative Site 110, Woodville South, South Australia
  - ACW Investigative Site 115, Carlton, Victoria
  - ACW Investigative Site 101, Ivanhoe, Victoria
  - ACW Investigative Site 108, Malvern, Victoria
  - ACW Investigative Site 112, Parkville, Victoria
  - ACW Investigative Site 104, Nedlands, Western Australia
  - ACW Investigative Site 109, West Perth, Western Australia